CLINICAL TRIAL: NCT04416711
Title: Reducing Alcohol-Related Sexual Risk Behavior
Brief Title: Alcohol And Sexual Risk Behavior
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Iowa (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA02771301A1
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Sexually Aggressive Behavior; Risky Sexual Behavior; Heavy Episodic Drinking
Keywords: Personalized Feedback; Cognitive Skills Training; Sexually Aggressive Behavior; Risky Sexual Behavior; Heavy Episodic Drinking

STUDY DESIGN:
Intervention Model Description: This two-site prevention trial will be conducted at Arizona State University (ASU) and the University of Iowa (Iowa). Participants will be 190 college men aged 18-19 (50% at each site). Scientific rigor will be ensured by (a) examining the feasibility of the intervention components in Phase I (n = 10); (b) evaluating the acceptability and preliminary efficacy of the intervention components in a Phase II open trial (n = 40); and (c) conducting a small randomized controlled trial (RCT; n = 140) in which participants will be randomly assigned (stratified by rape-supportive attitudes, frequency of HED, and frequency of sexual behavior) to either the treatment or services as usual (Phase III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services As Usual (Active Comparator): Participants assigned to the SAU condition will receive services as usual at their university, which include required programming related to heavy episodic drinking and sexually aggressive behavior either online or through new-student orientation.
  Interventions: Other: Services As Usual
- Personalized Feedback and Cognitive Training (Experimental): The prevention program will target heavy episodic drinking, sexually aggressive behavior, and risky sexual behavior through 2 sessions that integrate personalized feedback and cognitive training components.
  Interventions: Behavioral: Personalized Feedback; Behavioral: Cognitive Skills Training

INTERVENTIONS:
Behavioral: Personalized Feedback — The personalized feedback consists of four components: normative feedback, risk/protective feedback, decisional balance/goal setting, and protective strategy review. Personalized feedback targets include readiness to change, perceptions of risk, and misperceptions of peer attitudes/behaviors.
  Arms: Personalized Feedback and Cognitive Training
Behavioral: Cognitive Skills Training — We will address three cognitive targets: focus on affective cues, focus on non-affective cues, and over-perception of sexual interest. The first module targets enhanced focus on women's affective cues and reduced over-perception of sexual interest. We will introduce the role of men's sexual-perception skills in satisfying social and sexual interactions with women, as well as problematic sexual behavior including RSB and SAB. Next, we will instruct participants that affective information is the best-available nonverbal information about how a woman is feeling about a specific man. This instruction will focus on distinguishing four primary dating relevant cues: sexual-interest, friendliness, sadness, and rejection. More detailed focus on each cue will emphasize the increased difficulty of reading these cues with a new partner and under the influence of alcohol and sexual arousal, as well as the importance of checking verbally on assumptions about a woman's current sexual interest.
  Arms: Personalized Feedback and Cognitive Training
Other: Services As Usual — These participants will receive services as usual
  Arms: Services As Usual

SUMMARY:
The current study proposes to develop, refine, and conduct a preliminary randomized controlled trial (RCT) of an innovative prevention program that is the first to (a) simultaneously target heavy episodic drinking (HED), sexually aggressive behavior (SAB), and risky sexual behavior (RSB) among college men; (b) integrate personalized feedback and cognitive training strategies; and (c) target the five major modifiable risk factors for SAB: HED, impersonal sex, misperceptions of sexual interest, rape-supportive attitudes, and peer influence. The program will be computer-delivered as this approach is well received by college students.

DETAILED DESCRIPTION:
The study will include three phases (pilot feasibility n=10; pilot acceptability/efficacy n=40; RCT n=140), with 190 men at risk for HED, RSB, and SAB. Participants in the RCT will be randomly assigned to either the computer-based program or services as usual at 2 large public universities in the midwest and southwest U.S. The three study phases will address the following aims:

AIM ONE: Examine the feasibility of the computer administered personalized feedback and cognitive training approach (Phase I; n=10), and the acceptability and efficacy of individual intervention components based on skills assessments and interviews at 1-month follow-up (Phase II; n=40). Data from Phases I and II will be used to modify and streamline the intervention prior to the RCT (Phase III).

AIM TWO: In an RCT (n=140), evaluate whether the prevention program impacts cognitive training and personalized feedback targets at 1-month follow-up, relative to services as usual (SAU). Cognitive training targets include (a) enhanced focus on women's affect; (b) reduced focus on women's non-affective cues; and (c) correction of over-perceptions of women's sexual interest. Personalized feedback targets include (a) increased readiness to change; (b) increased perceptions of risk; and (c) reduced misperceptions of peer attitudes and behaviors.

AIM THREE: Evaluate whether the prevention program shows short-term effects on attitudinal (e.g., rape supportive and sociosexual attitudes) and behavioral outcomes (SAB, HED, and RSB) at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1) be male college students aged 18-19 at ASU or Iowa;
* 2) report at least one binge-drinking episode in the last month;
* 3) be unmarried and not engaged to be married;
* 4) be heterosexual or bisexual;
* 5) be dating or sexually active with women; and
* 6) be above the mean in rape supportive attitudes relative to 3000 college males in prior studies conducted at the two sites.

Exclusion Criteria:

* Do not meet the inclusion criteria

Ages: 18 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender eligibility is determined by both sex (male) at birth and identification (male).
Enrollment: 108 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
The Illinois Rape Myth Assessment | One month
  The Illinois Rape Myth Assessment - Short Form (IRMA-SF) will assess rape supportive attitudes (Payne, Lonsway, & Fitzgerald, 1999). Maximum values are 1 and maximum 7. Higher scores indicate more supportive attitudes.
Sociosexual Attitudes | One month
  Sociosexual attitudes will be assessed using 15 items from Bailey et al. (2000). This is not a validated scale but rather several items from past research. The scale ranges from 1 to 5, with higher scores being stronger attitudes.
Alcohol Use Disorder Identification Test | One month
  Heavy drinking will be assessed using the AUDIT. Specifically, one item asks about frequency of alcohol use, one item asks about frequency of binge drinking, and one item asks about quantity of alcohol use. Higher scores mean more drinking.
Attraction To Sexual Aggression | One month
  Rape proclivity will be assessed using the Attraction to Sexual Aggression scale (Malamuth, 1989a; Malamuth, 1989b), where participants rate their likelihood of engaging in sexual aggresion from 0-100%. Higher percentage equals higher attraction to sexual aggression.

SECONDARY OUTCOMES:
Risky Sexual Behavior | One month
  Engagement in risky sexual behavior will be assessed using 8 items from Bailey et al. (2000). Similar to sociosexual attitudes, these are items from a past study. Responses range from 1 to 7, with higher values indicating more risky sexual behavior.
Sexual Experience Survey | One month
  Will be assessed using a total of 21 items primarily based on the Sexual Experience Survey - Short Form Perpetrator (Koss et al., 2006a; Koss et al., 2006b; Koss et al., 2007). We will add all items together. Responses range from 1 to 4, with higher values indicating more sexual aggression.

CONTACTS AND LOCATIONS:
Overall Officials: William Corbin, PhD, Principal Investigator — Arizona State University; Teresa Treat, PhD, Study Chair — University of Iowa; Katie Witkiewitz, PhD, Study Chair — University of New Mexico
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Per NOT-AA-19-020, this study will submit and share data with NIAAA Data Archive (NIAAADA), a data repository housed within the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be uploaded into the NIMH NDA every April and October. The data collection is proposed to last 2.5 years.
Access Criteria: Access to the data will be granted through the NIMH NDA.

REFERENCES:
- [Background] Bohner G, Siebler F, Schmelcher J. Social norms and the likelihood of raping: Perceived rape myth acceptance of others affects men's rape proclivity. Pers Soc Psychol Bull. 2006 Mar;32(3):286-97. doi: 10.1177/0146167205280912. PMID 16455857
- [Background] Malamuth, N.M. (1989a). The attraction to sexual aggression scale: Part One. The Journal of Sex Research, 26, 26-49.
- [Background] Malamuth, N.M. (1989b). The attraction to sexual aggression scale: Part Two. The Journal of Sex Research, 26, 324-354
- [Background] Bohner, G., Reinhard, M.A., Rutz, S., Sturm, S., Kerschbaum, B., & Effler, D. (1998). Rape myths as neutralizing cognitions: Evidence for a causal impact of anti-victim attitudes on men's self-reported likelihood of raping. European Journal of Social Psychology, 28, 257-268.
- [Background] Babor, T. F., de la Fuente, J. R., Saunders, J., & Grant, M. (1992). AUDIT. The Alcohol Use Disorders Identification Test. Guidelines for Use in Primary Health Care. Geneva, Switzerland: World Health Organization.
- [Background] Sobell, L. C., & Sobell, M. B. (1992). Timeline Follow-back: A technique for assessing self-reported ethanol consumption. In J. Allen & R. Z. Litten (Eds.), Measuring Alcohol Consumption: Psychosocial and Biological Methods (pp. 41-72). Totowa, NJ: Humana Press.
- [Background] Kahler CW, Hustad J, Barnett NP, Strong DR, Borsari B. Validation of the 30-day version of the Brief Young Adult Alcohol Consequences Questionnaire for use in longitudinal studies. J Stud Alcohol Drugs. 2008 Jul;69(4):611-5. doi: 10.15288/jsad.2008.69.611. PMID 18612578
- [Background] Bailey JM, Kirk KM, Zhu G, Dunne MP, Martin NG. Do individual differences in sociosexuality represent genetic or environmentally contingent strategies? Evidence from the Australian twin registry. J Pers Soc Psychol. 2000 Mar;78(3):537-45. doi: 10.1037//0022-3514.78.3.537. PMID 10743879
- [Background] Larimer ME, Cronce JM. Identification, prevention, and treatment revisited: individual-focused college drinking prevention strategies 1999-2006. Addict Behav. 2007 Nov;32(11):2439-68. doi: 10.1016/j.addbeh.2007.05.006. Epub 2007 May 17. PMID 17604915
- [Background] Wood MD, Read JP, Palfai TP, Stevenson JF. Social influence processes and college student drinking: the mediational role of alcohol outcome expectancies. J Stud Alcohol. 2001 Jan;62(1):32-43. doi: 10.15288/jsa.2001.62.32. PMID 11271962
- [Background] Koss, M. P., Abbey, A., Campbell, R., Cook, S., Norris, J., Testa, M., Ullman, S., West, C., & White, J. (2006a). The Sexual Experiences Short Form Perpetration (SES-SFP). Tucson, AZ: University of Arizona.
- [Background] Koss, M. P. Abbey, A., Campbell, R., Cook, S., Norris, J., Testa, M., Ullman, S., West, C., & White, J. (2006b). The Sexual Experiences Long Form Perpetration (SES-LFP). Tucson, AZ: University of Arizona.
- [Background] Koss, M. P., Abbey, A., Campbell, R., Cook, S; Norris, J., Testa, C., Ullman, S., West, C., & White, J. (2007). Revising the SES: A collaborative process to improve assessment of sexual aggression and victimization. Psychology of Women Quarterly, 31, 357-370